CLINICAL TRIAL: NCT06167317
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GS-0201 as Monotherapy and in Combination in Adults With Advanced Solid Tumors
Brief Title: Study of GS-0201 Alone and in Combination in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-686-6854
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: GS-0201 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of GS-0201 monotherapy, until disease progression, or until the participant meets other study drug discontinuation criteria as specified in protocol or up to 105 weeks, whichever occurs first.
  Interventions: Drug: GS-0201
- Part B: Cohort B1: GS-0201 Monotherapy Dose Expansion (Experimental): Participants with selected indications will receive GS-0201 monotherapy at the recommended dose for expansion.
  Interventions: Drug: GS-0201
- Part B: Cohort B2: GS-0201 Monotherapy Dose Expansion (Experimental): Participants with selected indications not included in cohort B1 will receive GS-0201 monotherapy at the recommended dose for expansion.
  Interventions: Drug: GS-0201
- Part C: Dose Escalation: GS-0201 + Sacituzumab Govitecan (SG) (Experimental): Participants will receive escalating doses of GS-0201 in combination with SG, until disease progression, or until the participant meets other study drug discontinuation criteria as specified in protocol or up to 105 weeks, whichever occurs first.
  Interventions: Drug: GS-0201; Drug: Sacituzumab Govitecan
- Part D: Cohort D1: Dose Expansion: GS-0201 + SG (Experimental): Participants with confirmed unresectable locally advanced or metastatic triple negative breast cancer (mTNBC) will receive GS-0201 at the recommended Phase 2 dose (RP2D) in combination with SG.
  Interventions: Drug: GS-0201; Drug: Sacituzumab Govitecan
- Part D: Cohort D2: Dose Expansion: GS-0201 + SG (Experimental): Participants with confirmed unresectable locally advanced or metastatic HR+/HER2- breast cancer will receive GS-0201 at the recommended Phase 2 dose (RP2D) in combination with SG.
  Interventions: Drug: GS-0201; Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: GS-0201 — Pill administered orally
Drug: Sacituzumab Govitecan — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Part C: Dose Escalation: GS-0201 + Sacituzumab Govitecan (SG); Part D: Cohort D1: Dose Expansion: GS-0201 + SG; Part D: Cohort D2: Dose Expansion: GS-0201 + SG

SUMMARY:
The main goal of this first in human (FIH) study is to learn about the safety and dosing of GS-0201 when given alone or in combination with sacituzumab govitecan (SG) in participants with advanced solid tumors.

The primary objectives of this study are to:

* To assess the safety and tolerability of GS-0201 as monotherapy and in combination with SG in participants with selected advanced solid tumors
* To identify the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of GS-0201 as monotherapy and the MTD and/or the RP2D and dosing schedule of GS-0201 in combination with SG in participants with selected advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give written informed consent.
* Assigned female or male at birth, 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria by investigator assessment.
* Organ function requirements:

  * Adequate hematologic function
  * Adequate hepatic function
  * Creatinine clearance
  * Coagulation
* Tissue requirement:

  * Parts A, B, C, and D:

    * Pre-treatment tumor tissue is required.
  * Parts A and C backfill biopsy cohorts:

    * Participants must agree to fresh pre- and on-treatment biopsies.
* Participants assigned male at birth and participants assigned female at birth and of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Willing and able to comply with the requirements and restrictions in this protocol
* Part A (GS-0201 Monotherapy Dose Escalation) Inclusion Criteria:

  * Histologically/cytologically confirmed progressive/advanced solid tumors with selected molecular lesions.
  * Participants must have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit or have a contraindication to receive the therapy
* Part B (Dose Expansion) Inclusion Criteria:

  * Disease documented as:
  * Cohort B1:

    * Histologically or cytologically confirmed progressive/advanced selected solid tumor diagnoses harboring defined molecular lesions
    * Participants may potentially be required to forgo treatment with approved agent(s) to be able to participate in the study
  * Cohort B2:

    * Histologically or cytologically confirmed progressive/advanced solid tumor diagnoses harboring defined molecular lesions not included in Cohort B1
    * Participants must have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit or have a contraindication to receive the therapy
* Part C (Dose Escalation) Inclusion Criteria:

  * Histologically or cytologically confirmed unresectable locally advanced/metastatic selected solid tumors
* Part D (Dose Expansion) Inclusion Criteria:

  * Disease documented as:
  * Cohort D1:

    * Histologically or cytologically confirmed unresectable locally advanced or metastatic triple-negative breast cancer (mTNBC)
  * Cohort D2:

    * Histologically or cytologically confirmed unresectable locally advanced or metastatic HR+/HER2- (IHC 0, IHC 1+ or IHC 2+/ in situ hybridization (ISH-)) breast cancer.

Exclusion Criteria:

* Pregnant or lactating females
* Known hypersensitivity to any of the study drugs, its metabolites, or formulation excipients
* Requirement for ongoing therapy with or use of any prohibited medications described in the protocol
* Participants with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with findings suggestive of MDS/AML
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of GS-0201
* The therapies listed below within the specified timeframe:

  * Major surgery (excluding minor procedures, eg, placement of vascular access, gastrointestinal/biliary stent, biopsy) < 4 weeks prior to planned Cycle 1 Day 1
  * Immunotherapy or biologic therapy < 21 days prior to planned Cycle 1 Day 1
  * Chemotherapy < 14 days prior to planned Cycle 1 Day 1, or < 42 days for mitomycin or nitrosoureas
  * Targeted small molecule therapy < 14 days prior to planned Cycle 1 Day 1
  * Receipt of experimental therapy within 21 days or 5 experimental treatment half-lives (whichever is longer) prior to planned Cycle 1 Day 1
  * Hormonal or other adjunctive therapy for cancers other than the cancer under evaluation in this study that started < 14 days prior to planned Cycle 1 Day 1 are not permitted. Hormonal therapy, bisphosphonates, somatostatin analogues, and leuprolide are permitted if started ≥ 14 days prior to planned Cycle 1 Day 1
  * Radiotherapy within 2 weeks prior to planned Cycle 1 Day 1 and the radiation is not administered to a target lesion
  * Any prior allogeneic tissue/solid organ transplantation, including allogeneic hematopoietic stem cell transplantation. Participants with a history of autologous hematopoietic stem cell transplantation are also excluded
* Have not recovered (ie, Grade 1 or lower) from AEs due to a previously administered agent
* Prior treatment with approved or experimental prohibited agents as detailed in the protocol.
* Diagnosis of immunodeficiency, either primary or acquired, or requires systemic corticosteroids (> 10 mg of prednisone daily, or equivalent). However, replacement doses, topical, ophthalmologic, and inhalational steroids are permitted
* Have an active second malignancy
* Have known active central nervous system (CNS) metastases
* Participants with carcinomatous meningitis or primary CNS tumors are excluded regardless of clinical stability
* Meet any of the following criteria for cardiac disease:

  * Myocardial infarction or unstable angina pectoris within 6 months of enrollment
  * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication)
  * QT interval > 470 msec
  * New York Heart Association Class III or greater congestive heart failure or known left ventricular ejection fraction less than 40%
* Meet any of the following infectious criteria:

  * Have active serious infection requiring antimicrobials
  * Have active hepatitis B virus (HBV) or hepatitis C virus (HCV), or HIV. In participants with a history of HBV or HCV, participants with detectable viral loads will be excluded
  * Participants who test positive for hepatitis B surface antigen. Participants who test positive for hepatitis B core antibody are eligible with a negative HBV DNA by quantitative Polymerase chain reaction (PCR)
  * Participants who test positive for HCV antibody. Participants who test positive for HCV antibody are eligible with a negative HCV RNA by quantitative PCR
  * Participants who test positive for HIV antibody
* History of pneumonitis requiring treatment with corticosteroids, interstitial lung disease, or radiation pneumonitis requiring steroids
* Symptomatic ascites or pleural effusion
* Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the participant's participation in the study
* Use of any live vaccines against infectious diseases within 4 weeks (28 days) of initiation of study drug(s) (inactivated, viral vector vaccines, and messenger RNA (mRNA) vaccines are allowed; seasonal vaccines should be up to date prior to planned Cycle 1 Day 1)
* Parts C (Dose Escalation) and D (Dose Expansion): Combination Cohorts:

  * Participants with active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease) and participants with a history of bowel obstruction or gastrointestinal perforation within 6 months prior to planned Cycle 1 Day 1
  * Participants who previously received topoisomerase 1 inhibitors or antibody-drug conjugates containing a topoisomerase 1 inhibitor
  * Known severe intolerance or life-threatening hypersensitivity reactions to humanized monoclonal antibodies or intravenous (IV) immunoglobulin preparations; any history of anaphylaxis; history of human anti-human antibody response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The Number of Participants with Dose Limiting Toxicities (DLTs) During Dose Escalation | First dose up to 30 days post last dose (Up to approximately 109 weeks).
  DLTs are defined as any of the following treatment-emergent adverse events (AEs) regardless of attribution (graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0), unless clearly related to an underlying disease or extraneous causes, with onset within the DLT-evaluation period for the corresponding dose.
The Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose up to 30 days post last dose (Up to approximately 109 weeks).
The Incidence of Laboratory Abnormalities | First dose up to 30 days post last dose (Up to approximately 109 weeks).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Area Under the Concentration (AUC)0-24 of GS-0201 | Predose and postdose up to end of treatment (up to 105 weeks)
  AUC0-24 is defined as the concentration of drug over time between time 0 and time 24 hours.
PK Parameter: Cmax of GS-0201 | Predose and postdose up to end of treatment (up to 105 weeks)
  Cmax is defined as the maximum observed drug concentration.
PK Parameter: Tmax of GS-0201 | Predose and postdose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed concentration.
PK Parameter: AUC0-168 of SG (Parts C and D only) | Predose and postdose up to end of treatment (up to 105 weeks)
  AUC0-168 is defined as the concentration of drug over time between time 0 and time 168 hours.
PK Parameter: Cmax of SG (Parts C and D only) | Predose and postdose up to end of treatment (up to 105 weeks)
  Cmax is defined as the maximum observed drug concentration.
PK Parameter: Tmax of SG (Parts C and D only) | Predose and postdose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed concentration.
GS-0201 Plasma Concentrations | Predose and postdose up to end of treatment (up to 105 weeks)
Sacituzumab Govitecan (SG) Serum Concentrations (Parts C and D only) | Predose and postdose up to end of treatment (up to 105 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NEXT Austin, Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Dallas, Irving, Texas
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06167317